CLINICAL TRIAL: NCT04874103
Title: Endoscopic Ultrasound-guided Gallbladder Drainage in High Surgical Risk Patients With Acute Cholecystitis: Prospective Evaluation of the Hong Kong Follow up Protocol
Brief Title: Hong Kong Follow up Protocol After EUS Gallbladder Drainage for Acute Cholecistitis
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Other Study IDs: EUS-GBD Hong Kong
Record Dates: First submitted 2021-04-27; First posted 2021-05-05 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis, Acute
Keywords: endoscopic ultrasound; eus; acute cholecistitis; gallbladder drainage
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUS guided gallbladder drainage and cholecystoscopy: EUS-GBD will be performed using LAMS (such as Hot-AxiosTM device). A 10mm x 10mm stent system will be used if the largest gallstone is smaller than 10mm in size and a 15 x 10mm stent will be used if the largest gallstone is larger than 10mm.
  Colecystoscopy will be subsequently performed after at least 2 weeks using standard or therapeutic gastroscope. Lithotripsy will be performed using mechanical lithotripsy or laser lithotripsy.

SUMMARY:
This study evaluates the long-term safety and efficacy of the Hong Kong follow up protocol in patients who will undergo drainage of the gallbladder under endoultrasonography (EUS) guidance in patients with acute cholecistitis not suitable for surgery.

DETAILED DESCRIPTION:
Acute cholecystitis is a common surgical condition. However, in elderly patients or patients with significant comorbidity, emergency laparoscopic cholecystectomy can be associated with significant risk of morbidities. Thus, in these patients, percutaneous cholecystostomy (PC) could be employed for drainage of the gallbladder. However, complications including intrahepatic hemorrhage, pneumothorax, biliary peritonitis and pneumonia have been reported in a mean of 6.2% of patients (range 0-25%). Furthermore, PC has several other disadvantages including risk of bile leakage, recurrent cholecystitis, inadvertent tube removal and migration (0-25%), necessitating repeated procedures. In order to avoid nuisances associated with PC, studies looking at potential ways to achieve endoscopic gallbladder drainage have been performed. On the other hand, EUS-guided transmural drainage procedures are increasingly performed for management of a variety of conditions and has also been described for drainage of the gallbladder in patients that are not fit for surgery since 2007. Recently, a lumen-apposing metal stent (LAMS) has become available which allows easier deployement of the stent. A 9.8mm gastroscope or a 5mm ultrathin nasal endoscope can pass through the lumen of the stent and enter the gallbladder for stone removal or other interventions A recent study group from Hong Kong promoted a specific follow up for EUS guided gallbaldder drainage patients who underwent a follow-up cholecystoscopy after the procedure to check for clearance of stones. In patients with stones that were too large to pass out spontaneously, basket mechanical lithotripsy was employed to break down the stones, followed by laser lithotripsy if the latter was not successful. No data on the safety and efficacy of the Hong Kong follow up protocol in patients who underwent EGBD using LAMS coming from countries other than Asian are available, in which differences in etiological and pathogenic factors might not required such an intensive follow up protocol. To explore this important question we have designed a study aimed at evaluating the long-term safety and efficacy of the Hong Kong follow up protocol in patients undergoing EGBD performed using LAMS.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with acute cholechystitis unsuitable for surgery
* age ≥ 18 years old
* Written informed consent from patient or guardian who is able to understand the nature and possible consequences of the study

Exclusion Criteria:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients with suspected gangrene or perforation of the gallbladder
* Patients diagnosed with concomitant liver abscess or pancreatitis (defined as elevated serum amylase more than three times the upper limit of normal)
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Patients with liver cirrhosis, portal hypertension and/or gastric varices
* Abnormal coagulation (INR > 1.5 and/or platelets < 50.000/mm3)
* Contraindication to perform endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns consecutive patients undergoing EGBD using LAMS as per decision of the on call surgeons of the Emergency Surgery Department with diagnosis of acute cholecystitis, who are unsuitable for early laparoscopic cholecystectomy due to poor premorbid conditions
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events after EUS gallbladder drainage and cholecystoscopy | From date of treatment every 2-3 months, assessed until death or up to 2 years
  Percentage adverse events after the procedures. Adverse events will be considered major if they prevent completion of the scheduled procedure and/or resulted in prolongation of hospital stay, another therapeutic procedure (needing sedation/anesthesia), or subsequent medical consultation. Any potential adverse event such as pancreatitis, burns of the gastric or duodenal walls, bowel injury, or peritonitis will be recorded and graded according to the above-mentioned classification.
Incidence of recurrent acute cholecystitis after EUS-GBD and cholecystoscopy | From date of treatment, every 2-3 months, assessed until death or up to 2 years
  Percentage of patients with recurrent acute cholecystitis symptoms after EUS-GBD and cholecystoscopy with residual stone removal if present after resolution of the index episode.

SECONDARY OUTCOMES:
Incidence of patients with resolution of acute cholecystitis symptoms after EUS-GBD | Within 96 hours after procedure
  Percetange of patients achieving acute cholecystitis symptoms resolution after EUS-GBD demonstrated by normalization of clinical parameters of acute cholecystitis within 96 hours. Clinical parameters reported are abdominal pain evaluated by the patients on a 10-point visual analogue scale, temperature, white blood cell count and serum C-reactive protein concentration.
Need for advaced gallbladder interventions | From date of treatment, every 2-3 months, assessed until death or up to 2 years
  Number of patients who will require more advanced gallbladder interventions during follow up such as colecystoscopy lithotripsy will be assessed by the numebr of patients who will require such treatments.
Need for ERCP | From date of treatment, every 2-3 months, assessed until death or up to 2 years
  rate of patients who will require ERCP due to stones migration during colecystoscopy will be assessed by the number of patients who will require such intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, MD, Phd, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Universita' Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SS, Park DH, Hwang CY, Ahn CS, Lee TY, Seo DW, Lee SK, Kim MW. EUS-guided transmural cholecystostomy as rescue management for acute cholecystitis in elderly or high-risk patients: a prospective feasibility study. Gastrointest Endosc. 2007 Nov;66(5):1008-12. doi: 10.1016/j.gie.2007.03.1080. Epub 2007 Sep 4. PMID 17767933
- [Background] Keus F, Gooszen HG, van Laarhoven CJ. Open, small-incision, or laparoscopic cholecystectomy for patients with symptomatic cholecystolithiasis. An overview of Cochrane Hepato-Biliary Group reviews. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD008318. doi: 10.1002/14651858.CD008318. PMID 20091665
- [Background] Kwan V, Eisendrath P, Antaki F, Le Moine O, Deviere J. EUS-guided cholecystenterostomy: a new technique (with videos). Gastrointest Endosc. 2007 Sep;66(3):582-6. doi: 10.1016/j.gie.2007.02.065. PMID 17725950
- [Background] Teoh AYB, Serna C, Penas I, Chong CCN, Perez-Miranda M, Ng EKW, Lau JYW. Endoscopic ultrasound-guided gallbladder drainage reduces adverse events compared with percutaneous cholecystostomy in patients who are unfit for cholecystectomy. Endoscopy. 2017 Feb;49(2):130-138. doi: 10.1055/s-0042-119036. Epub 2016 Nov 22. PMID 27875855